CLINICAL TRIAL: NCT04588844
Title: Effect of Polyethylene Glycol Recombinant Human Growth Hormone Injection on the IVF/ICSI Outcome of Patients With Poor Ovarian Reserve
Brief Title: Effect of Growth Hormone Injection on the IVF/ICSI Outcome of Patients With Poor Ovarian Reserve.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shandong University (Other)
Collaborators: RenJi Hospital (Other); The Second Hospital of Hebei Medical University (Other)
Responsible Party: Principal Investigator, Chen Zi-Jiang, Professor, Shandong University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PEG-rhGH
Record Dates: First submitted 2020-10-09; First posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Poor Ovarian Reserve

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Growth Hormone group (Experimental): Growth Hormone pretreatment for 6 weeks before ovarian stimulation
  Interventions: Drug: Polyethylene Glycol Recombinant Human Somatropin
- Control group (No Intervention): No pretreatment before ovarian stimulation

INTERVENTIONS:
Drug: Polyethylene Glycol Recombinant Human Somatropin — Polyethylene glycol recombinant human somatropin will be injected weekly (3mg/per week) from the beginning of preceding menstruation cycle until the day of ovum pickup.
  Arms: Growth Hormone group

SUMMARY:
Declined fertility and ovarian reserve in older women are associated with lower density of Growth hormone (GH) receptors and dysregulation in GH secretion. GH can regulate the expression of growth hormone receptor and strengthen the function of mitochondria, which could improve the quality of the female oocyte. In this study, a prospective randomized control will be conducted to explore the effect of GH adjuvant therapy on clinical outcome of in vitro fertilization.

DETAILED DESCRIPTION:
Eligible subjects will be randomly assigned into either the study groups (receive somatropin co-treatment) or the control group (without sopmatropin treatment). Polyethylene glycol recombinant human somatropin will be injected weekly (3mg/per week) for approximately 6 weeks, i.e. from the beginning of preceding menstruation cycle until the day of ovum pickup. Both groups will receive a similar common protocol for ovarian stimulation. In vitro fertilization with or without intracytoplasmic sperm injection will be performed according to semen parameters. All embryos will undergo culture for blastocyst and the obtained blastocysts will be vitrified for deferred frozen embryo transfer. The Blastocyst formation rate will be the primary outcome measure.

ELIGIBILITY:
Inclusion Criteria:

* 1)Married women between 35-40 years old; 2) serum AMH< 1.2ng/ml, and basal FSH<20IU/L during the screening period or within 6 months; 3) 18kg/m2≤BMI<30kg/m2; 4) Previous ART cycles <3.

Exclusion Criteria:

* 1）Gynecological diseases that affect pregnancy outcomes, such as submucous uterine myoma, intramural uterine myoma≥4cm, Ovarian cyst≥4cm, endometriosis, Uterine malformation, Tuberculosis of reproductive system; 2) Spontaneous abortion≥3 times; 3) Chromosomal abnormalities (except polymorphism) in one or both spouses; 4) Patients with well-defined and uncontrolled endocrine, metabolic, and adrenal diseases, such as diabetes, thyroid disease, Cushing's syndrome; 5) Patients with malignant tumors; 6) Previous use of somatropin products.

Ages: 35 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2022-03-20 (Estimated); Study Completion 2023-03-20 (Estimated)

PRIMARY OUTCOMES:
Blastocyst formation rate | One year
  the number of blastocyst/ the total number of embryos underwent blastocyst culture ×100%
Live birth rate | One year

SECONDARY OUTCOMES:
Number of retrieved oocytes | One year
Number of high-score embryos | One year
total amount of Gn used | One year
total days of Gn administration | One year
clinical pregnancy rate | One year
Ongoing pregnancy rate | One year
E2 levels on triggering day | One year
Endometrial thickness on triggering day | One year

IPD SHARING:
Plan to Share IPD: Yes
The study protocol and statistical analysis plan will be available online with publication. Data collected for the study, including specified data set and a data dictionary defining each field in the set, will be made available to others with publication.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After publication and for 1 year
Access Criteria: Investigators can request data sharing by contacting the email of the corresponding author. Our publication committee established for this trial will review and approve the request.